CLINICAL TRIAL: NCT03638583
Title: Alzheimer Prevention Trials (APT) Webstudy
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Brigham and Women's Hospital (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Paul S. Aisen, Professor, University of Southern California
Other Study IDs: HS-17-00746; R01AG053798 (NIH)
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Alzheimer's; Prevention; Web-Based
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of the Alzheimer Prevention Trials (APT) Webstudy is to accelerate enrollment for Alzheimer's disease (AD) clinical trials by identifying and tracking individuals who may be at higher risk for developing AD dementia.

DETAILED DESCRIPTION:
The APT Webstudy will use web-based cognitive testing and questionnaires to generate a risk score which will be used to identify individuals who may be at an increased risk for developing AD dementia.

Individuals who join the APT Webstudy will register at https://www.aptwebstudy.org/, sign an electronic informed consent form (ICF), provide basic demographic information and participate in web-based cognitive testing. Participants will return the APT Webstudy quarterly (every 3 months) to complete the cognitive testing again.

Based on the risk score and changes identified in the cognitive testing results, participants will be invited to visit a partnering clinical trial site for an in-person visit with biomarker testing and clinical assessment.

The combined results of the web-based assessments, with the biomarker and clinical assessments, will allow an adaptive statistical algorithm to improve the selection of those at highest risk for developing AD.

To Join the APT Webstudy, please visit https://www.aptwebstudy.org/.

ELIGIBILITY:
Inclusion Criteria:

* male or female at least 50 years of age
* no evidence of dementia
* willing to participate in remote longitudinal cognitive testing and possible referral for biomarker assessment based on risk

Exclusion Criteria:

* N/A. Anyone can register for the APT Webstudy, however, only individuals identified using the risk algorithm will be referred for in-person biomarker assessments.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anyone who meets entry criteria is eligible to join the Webstudy. We anticipate 200,000 individuals will join.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Enrollment into Alzheimer's prevention research studies | 5 years

SECONDARY OUTCOMES:
Referral into prevention research studies | 5 years
Number of individuals enrolled into Alzheimer's prevention studies | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Aisen, MD, Principal Investigator — USC ATRI; Reisa Sperling, MD, Principal Investigator — Brigham and Women's Hospital; Jeffrey Cummings, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Https://Www.Aptwebstudy.Org, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No